CLINICAL TRIAL: NCT00248092
Title: A Double-Blind, Randomized, Placebo and Active-Controlled, Six-Period Crossover Study to Evaluate the Likeability, Safety, and Abuse Liability of NRP104 in Healthy Adult Volunteers With Histories of Stimulant Abuse
Brief Title: Study to Evaluate the Likeability, Safety, and Abuse Potential of NRP 104 in Adults With Histories of Stimulant Abuse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRP104.A03
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Amphetamine-Related Disorders; Substance-Related Disorders
Keywords: d-Amphetamine; Diethylpropion; Diethylpropion Hydrochloride; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders with Hyperactivity; Attention Deficit Hyperactivity Disorders; Amphetamine Abuse; Amphetamine Dependence; Amphetamine Addiction; Amphetamine Users; Drug Abuse; Drug Addiction; Drug Dependence; Drug Habituation; Drug Use Disorders; Substance Abuse; Substance Dependence; Substance Use Disorders; Drug Usage; Substance Addiction
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Amphetamine-Related Disorders; Substance-Related Disorders | interventions — Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: NRP104

SUMMARY:
This research is being done to evaluate if NRP104 is a safe drug. The other purpose is to learn if NRP104 produces a high and any other effects like amphetamine and other stimulant drugs that are abused. This information will give some indication if NRP104 can be abused. NRP104 is an investigational drug. This means that it has not been approved by the U.S. Food and Drug Administration (FDA). Healthy people, between the ages of 18 and 55 with histories of substance abuse that include stimulant drugs, may join. Amphetamines are drugs that are used most often to treat attention deficit hyperactivity disorder (ADHD) in children, to treat narcolepsy (excessive sleepiness) and for weight loss.

DETAILED DESCRIPTION:
There is a need for a less abusable stimulant medication that can provide symptom control for children with ADHD as compared to the conventional stimulant products.

Currently, the top line amphetamine product Adderall XR(R) for the treatment of children with ADHD involves a once-a-day morning dosing of up to 30 mg per day per Adderall XR(R) Package Insert. Adderall XR(R) has potential for abuse and is hence is classified as a schedule II product.

As part of the development of NRP104 for treatment of children with ADHD, it is important to evaluate the abuse potential of NRP104 in comparison to immediate release d-amphetamine. A previous exploratory dose ranging study (NRP104.A01) with NRP104 demonstrated that doses of NRP104 up to 150 mg are safe and produce effects equal to or less than 40 mg of immediate release d-amphetamine. When compared with those of d-amphetamine, diethylproion produced effects qualitatively similar to those of d-amphetamine but were significantly less potent. Intravenous and subcutaneous routes diethylpropion was less potent as compared to oral route (Jasinski et al; 1974). This larger study is designed to compare the abuse potential of NRP104 with the Schedule II d-amphetamine sulfate and the Schedule IV diethylpropion hydrochloride. Data collected from this study will be used to evaluate the abuse potential of NRP104.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject is 18 to 55 years of age, inclusive.
* Except for women who are post menopausal or surgically sterile, all female subjects must have a negative urine pregnancy test at screening and at admission. They must abstain from sexual activity, or use acceptable contraceptives throughout the study, and for 30 days after the last dose of study drug. Acceptable contraceptives include double barrier method (such as condom with spermicidal gel or diaphragm with spermicidal gel), IUDs and hormonal contraceptives which must be pharmacologically effective prior to study drug exposure.
* Meet DSM-IV criteria for the diagnosis of substance abuse.
* Subject must be in good health and have venous access sufficient for blood collection, as determined by medical history, physical exam, and clinical labs.
* Agree to be admitted to the inpatient research unit for a minimum of 14 days, and will be able to complete all protocol-specified assessments.
* Able to understand that they can withdraw from the study at any time.
* Minimum reading level of Grade Six as determined by the REALM test, at the investigator's discretion.
* Subject must voluntarily consent to participate in this study.
* Able to swallow the study medication whole.

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, endocrine, oncologic, hematologic, neurologic, psychologic, immunologic or pulmonary disorders; or cardiovascular disease, tuberculosis, epilepsy, diabetes, psychosis, glaucoma, or any condition which in the opinion of the Investigator would jeopardize the safety of the subject or impact study results or prevent the subject from completing the study.
* Presence or history of any medically diagnosed, clinically significant Axis I psychiatric disorders other than substance abuse (including bipolar disorder, any psychotic disorder, and Tourette's disorder or family history of Tourette's).
* Serious suicidal risk determined by the investigator.
* Presence of a severe learning difficulty or mental retardation, or any condition that would interfere with participation or completion of the study.
* History of allergic or adverse response or hypersensitivity to d-amphetamine or NRP104.
* Participation in a previous clinical trial within 30 days prior to study initiation.
* Blood loss, donation of one pint or more, or plasma donation within 60 days prior to study initiation.
* Clinically significant abnormalities at screening or admission on results of ECG or lab tests, including lab deviations requiring acute medical intervention or further medical attention.
* Treated with a monoamine oxidase inhibitor, currently or within 13 days of initiation of the study medication.
* Require any of the following medications: clonidine or other alpha-2 adrenergic receptor agonists, tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs) theophylline, coumarin anticoagulants, or anticonvulsants; or have taken an SSRI in the 35 days before initiation of the study medication.
* Currently physically dependent on benzodiazepines as determined by clinical evaluation and/or urine drug screen at screening.
* Currently physically dependent on opiates as determined by naloxone challenge.
* Currently physically dependent on alcohol as determined by clinical evaluation or has a confirmed positive Breathalyzer test at screening or admission.
* Preexisting severe gastrointestinal narrowing.
* Use of any prescription medications (except birth control) within 14 days of admission, or will require any prescription medications, or any over-the-counter (OTC) medications (other than acetaminophen), or herbal supplements or vitamins during the study.
* Positive urine pregnancy test at screening or admission.
* Female subject is pregnant or lactating.
* Related to any person directly or indirectly involved with the conduct of the study or currently participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2006-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The difference in the time to maximum change from baseline in the Liking scale score (Question 2) from the Drug Rating Questionnaire - Subject (DRQS).

SECONDARY OUTCOMES:
Maximum Liking score (Question 2 from DRQS) change from baseline
Question 1 and 3 from the DRQS
Question 1, 2 and 3 from the Drug Rating Questionnaire- Observer (DRQO)
Subscale of the ARCI (MBG, Amphetamine, BG, LSD and PCAG) (subject)
Street Value assessment Questionnaire (subject)
Treatment Enjoyment assessment Questionnaire (TEAQ) (subject)
Safety
Adverse events, laboratory tests, physical examination, vital signs and ECG will be collected to
assess the safety and tolerability of NRP104.

CONTACTS AND LOCATIONS:
Overall Officials: Donald R. Jasinski, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Clinical Studies Program, Baltimore, Maryland, United States